CLINICAL TRIAL: NCT02226848
Title: Effect of Administration of Recombinant Erythropoietin on Numbers of Circulating Endothelial Progenitor Cells in Patients With Persistent Symptoms During the Subacute Period After TBI
Brief Title: Effect of Recombinant Erythropoietin on Numbers of Circulating Endothelial Progenitor Cells in People With Persistent Symptoms During the Subacute Period After Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 140174; 14-N-0174
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-05-31

CONDITIONS: Traumatic Brain Injury
Keywords: Endothelial Progenitor Cells; Angiogenesis; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

INTERVENTIONS:
Drug: Erythropoeitin

SUMMARY:
Background:

- Traumatic brain injury (TBI) injures blood vessels in the brain. Endothelial progenitor cells (EPCs) help the body form new blood vessels. The drug erythropoietin (EPO) helps the body make more blood cells and might help make blood vessels. Researchers want to see if EPO helps people with TBI.

Objective:

- To see whether erythropoietin increases the number of endothelial progenitor cells circulating in the blood and changes reactivity of brain vessels.

Eligibility:

- Adults age 18 70 who had a TBI 3 7 days ago and still have symptoms.

Design:

* Participants will be screened with medical history and blood tests. Vital signs will be taken.
* Visit 1:
* Medical history, physical exam, and blood sample.
* Neuropsychological tests of memory, attention, and thinking. These include written and spoken questions, tests on paper or computer, and simple actions.
* Magnetic resonance imaging (MRI) scan with carbon dioxide. Participants will lie on a table that slides in and out of a metal cylinder. For part of the scan, participants will wear a breathing mask like a snorkel and wear a nose clip.
* Study drug or placebo injection under the skin of the arm, leg, or buttock.
* Visits 2, 3, and 4 will be 1 week apart.
* Blood sample.
* Review of TBI symptoms and any drug side effects.
* Study drug or placebo injection under the skin.
* Visit 5 will be 1 week after visit 4. Visit 6 will be 6 months after participants start the study.
* Blood sample.
* Review of TBI symptoms and any drug side effects.
* Neuropsychological tests.
* MRI with carbon dioxide.

DETAILED DESCRIPTION:
Objective

Traumatic brain injury (TBI) is the leading cause of death and disability in people under age 45 in industrialized countries 5;6. Significant numbers of US veterans from the wars in Iraq and Afghanistan return with TBI7. However, to date, there are no specific neuroprotective treatment options with proven clinical efficacy 8. Erythropoietin (EPO) is approved by the FDA to treat anemia and has comprehensive preclinical data supporting its neuroprotective and neuroregenerative efficacy following traumatic (TBI) and a wide range of other acquired brain insults. Injury to small and medium-sized cerebral blood vessels is a well recognized consequence of TBI. EPO increases production of endothelial progenitor cells (EPCs) 4;9 and promotes angiogenesis and neovascularization after TBI. EPO also promotes neurogenesis and improves functional recovery in animals after experimental stroke10-12 and TBI.13;14 Neovascularization is coupled with neurogenesis, and augmentation of both processes by EPO may result in lessened cognitive deficits. Neovascularization by EPO may prevent post-traumatic deficits in cerebrovascular reactivity (CVR), which can be measured noninvasively using magnetic resonance imaging (MRI).

This proposal is for a randomized, placebo-controlled pilot clinical trial designed to obtain data on the effects of EPO in humans with persistent post-concussive symptoms after TBI. The primary objective is to evaluate effect of 4 week administration of recombinant erythropoietin on numbers of circulating endothelial progenitor cells in patients with persistent symptoms during the subacute period after TBI. This information will guide the design of a future definitive study.

Study Population

The study population will include 30 males and females with persistent post-concussive symptoms continuing up to 7 days after TBI. Participants will be military service members or civilians presenting as outpatients for clinical management of TBI or post-concussive symptoms at the Center for Neuroscience and Regenerative Medicine (CNRM)-affiliated hospitals. These include the Walter Reed National Military Medical Center (WRNMMC), Suburban Hospital (SH), and Washington Hospital Center (WHC).

Design

Participants will be referred to the NIH Clinical Center (CC) from participating hospitals or will be recruited by advertisements through CNRM Recruitment core to receive EPO or placebo. Telephone screening will be carried out to determine tentative eligibility. At the baseline visit, participants will be screened, consented and randomized 2:1 to receive either EPO or placebo with a dose of 40,000 IU EPO subcutaneously (s.c.) (n=20) once weekly for 4 weeks or placebo (n=10). Each participant will have 6 outpatient visits (visits 1-6) performed at the NIH CC. Placebo or active drug will be administered s.c. based on the randomization at visits 1-4; blood will be collected for EPC assays and safety laboratory measurements during each visit. Brain MRI and neuropsychological tests will be performed during visit 1 (before administering EPO or placebo), and visit 5 (one week after final drug administration) and visit 6 (6 months after study enrollment).

Outcome Measures

Primary outcome:

1. . Effect of 4 weeks of EPO administration on numbers of circulating EPCs in patients with persistent symptoms during the subacute period after TBI (within subject comparison).

   Secondary outcomes:
2. . Comparison of the change of numbers of circulating EPC s between EPO and placebo groups.
3. . Effect of 4 weeks of EPO administration on MRI biomarkers of TBI recovery (such as CVR on hypercapnia and global and regional brain volumes by MRI).
4. . Effect of 4 weeks of EPO administration on plasma biomarkers of angiogenesis and inflammation, such as stem cell factor (SCF), vascular endothelial growth factor (VEGF), stromal-derived factor (SDF-1 ); and matrix metalloproteinase-9 (MMP-9).
5. . Effect of 4 weeks of placebo administration on numbers of circulating EPCs in patients with persistent symptoms during the subacute period after TBI.

   Tertiary outcome:
6. . Relationship between EPC levels at baseline and after 4 weeks and neuropsychological performance following TBI.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 - 70 years, inclusive
  2. History of having sustained a TBI greater than or equal to 3 days and less than or equal to 7 days prior to enrollment. This evidence will be any one of the following:

     1. GCS 3 - 12 on first presentation to medical attention
     2. Post-traumatic amnesia > 24 hours
     3. TBI-related abnormality on neuroimaging (either CT or MRI)
  3. Persistent post-concussive symptoms, according to the DSM-IV Research Criteria for Post- Concussional Disorder.

     1. Three of more of the following symptoms, which started shortly after the trauma and persist for at least up to the time of enrollment:

        * Fatigueability
        * Disordered sleep
        * Headache
        * Vertigo or dizziness
        * Irritability or aggression
        * Anxiety, depression, or affective instability
        * Changes in personality (e.g., social or sexual inappropriateness)
        * Apathy or lack of spontaneity
     2. Symptoms had their onset after trauma, or there is a significant worsening or preexisting symptoms after trauma.
  4. Ability to read, write, and speak English
  5. Ability to give consent by the participant himself
  6. Willingness of women of childbearing potential to use effective contraception during this study and until 2 weeks after they have completed the study drug (EPO or placebo).

Effective methods of contraception for this study include:

* hormonal contraception (birth control pills, injected hormones or vaginal ring),
* intrauterine device,
* barrier methods (condom or diaphragm) combined with spermicide,
* surgical sterilization (hysterectomy, tubal ligation), or vasectomy in a partner.

EXCLUSION CRITERIA:

1. Contraindication to EPO therapy:

   1. Known allergy to EPO, hypersensitivity to mammalian cell-derived products, or hypersensitivity to albumin
   2. Serum hemoglobin > 16 g/dL in a male patient or > 14 g/dL in a female patient; or a platelet count > 400,000/mm3 or serum hemoglobin < 10 g/dL in either a male or female patient
   3. liver or kidney disease; the former will be operationally defined as a serum bilirubin > 4 mg/dL, alkaline phosphatase (AP) > 250 U/L, aspartate aminotransferase (SGOT, AST) > 150 U/L, alanine aminotransferase (SGPT, ALT) >150 U/L, or Moderately decreased GFR 30-59 ml/min/1.73m2
   4. Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female of childbearing potential
2. Use of EPO one month prior to the randomization
3. Suspicion of a coagulation disorder associated with bleeding (PTT>45 or INR>1.7, spontaneously out of normal range)
4. Pre-existing and active major disabling psychiatric disorder (e.g., schizophrenia or bipolar disorder), or other neurological disease (epilepsy, multiple sclerosis, developmental disorder) not related to TBI
5. History of heart disease or heart attack, congestive heart failure, stroke, venous thromboembolism.
6. History of disorders that predispose to coagulation (e.g. polycythemia vera, essential thrombocytosis, or thrombotic thrombocytopenic purpura).
7. Uncontrolled hypertension, defined as above 140/90 mm Hg in three measurements in two separate visits despite antihypertensive therapy. Antihypertensive therapy is allowed, including agents such as thiazide diuretics, ACE inhibitors, beta-blockers, calcium channel blockers, alpha-blockers, or a centrally acting alpha agonists.
8. Known malignant conditions, e.g., melanoma, breast, brain, lung tumor or prostate cancer
9. Terminal medical diagnosis consistent with survival < 1 year
10. Planned surgical procedure during duration of the study (if emergency surgery needed, EPO administration will be stopped, but the patient will remain in the study according to the intention to treat principles).
11. Current use of Coumadin or other blood thinners (e.g. Pradaxa, Heparin, Lovenox)

    ASA, Plavix or Aggrenox are not a contraindication
12. Any history of previous deep venous thrombosis (DVT), pulmonary embolization (PE), or other thromboembolic event
13. Current participation in other interventional clinical trial
14. Current use of iron supplements
15. Evidence of penetrating brain injury
16. Contraindication to MRI scanning
17. No adherence to use of effective method of contraception for females of childbearing potential for time from enrollment to the study until 2 weeks after completion of the study drug (EPO or placebo)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08-15; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Effect of 4 weeks of EPO administration on numbers of circulating EPCs in patients with persistent symptons during the subacute period after TBI. | 4 weeks

SECONDARY OUTCOMES:
Safety of 4 weeks of EPO administration to TBI participants | 4 weeks
Effect of 4 weeks of EPO administration on MRI biomarkers of TBI recovery | 4 weeks
Effect of 4 weeks of EPO administration on biomarkers | 4 weeks
Relationship between EPC levels at baseline after 4 weeks and neuropsychological performance following TBI. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)